CLINICAL TRIAL: NCT01939834
Title: Early Feasibility Study of Adaptive Advisory/Automated (AAA) Control of Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subjects preferred the 5 night overnight system in terms of ease of use.
Sponsor: Sue Brown (Other)
Collaborators: DexCom, Inc. (Industry); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor-Investigator, Sue Brown, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 16930
Record Dates: First submitted 2013-08-14; First posted 2013-09-11 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Artificial Pancreas; Diabetes Assistant (DiAs); Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Overnight CLC followed by SAP (Experimental): Throughout the trial, participants wore a study CGM. Participants spent 5 nights in a supervised outpatient setting using closed-loop control (CLC) system running on DiAs from 23:00 to 07:00. The participants then subsequently had a week at home in which they wore either their personal pump (UVA) or the study pump (Italy) along with a continuous glucose monitor without running in any specialized mathematical equations (sensor-augmented pump therapy or SAP). Four fingersticks completed each day and carbohydrates will be recorded in bolus calculator of their insulin pump prior to each meal.
  Interventions: Device: Overnight CLC; Device: Sensor-Augmented Pump Therapy (SAP)
- SAP followed by Overnight CLC (Experimental): Throughout the trial, participants wore a study CGM. Participants in this arm spent a week had a week at home in which they wore either their personal pump (UVA) or the study pump (Italy) along with a continuous glucose monitor without running in any specialized mathematical equations (sensor-augmented pump therapy or SAP). They subsequently spent 5 nights in a supervised outpatient setting using closed-loop control (CLC) system running on DiAs from 23:00 to 07:00. Four fingersticks completed each day and carbohydrates will be recorded in bolus calculator of their insulin pump prior to each meal.
  Interventions: Device: Overnight CLC; Device: Sensor-Augmented Pump Therapy (SAP)

INTERVENTIONS:
Device: Overnight CLC — Overnight Closed-Loop Control (CLC) is run on the DiAs which is a medical platform that uses a smart-phone to connect to a continuous glucose sensor to insulin pump. The cell phone runs the CLC and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range.
Device: Sensor-Augmented Pump Therapy (SAP) — The subject will be on their home insulin pump (UVA) or study pump (Italy) and using a CGM per their usual care.

SUMMARY:
The purpose of this study is to use an Advisory/Automated Adaptive (AAA) or Closed-Loop Control (CLC) system for insulin delivery in adults with Type 1 Diabetes (T1DM) in an outpatient setting to evaluate the system's ability to significantly improve blood glucose levels. A component of this study evaluated AAA or CLC Control overnight only in 5 consecutive overnights in a cross-over trial with sensor-augmented pump therapy occurring prior to or following CLC overnight. Another component of this study planned evaluating if the AAA Control system run on the Diabetes Assistant (DiAs) system can prevent hypoglycemia during and following exercise more efficiently during a 40 hour trial this part of the trial was not conducted due to a preference for overnight only configuration in pilot testing. This protocol represents a culmination of prior clinical trials in development of this AAA system and benefits from the synthesis of those components.

DETAILED DESCRIPTION:
The primary goal of this study is to test an Advisory/Automated Adaptive (AAA) or CLC Control system, which includes three interacting control modules:

* Module 1 - Automated Safety Supervision (SSM) responsible for prevention of hypoglycemia, which can be adapted (individualized) with prior data for each subject;
* Module 2 - Advisory Module (AM) responsible for pre-meal boluses and postprandial corrections, which can be adapted (individualized) with prior data for each subject;
* Module 3 -- Automated Basal Rate Module (BRM) responsible for augmentation of basal rate to compensate for changes in insulin sensitivity, particularly overnight (e.g. dawn phenomenon), which can be adapted with prior data for each subject.

Daytime control (40hour studies) includes all 3 modules (n=36 were not recruited). Overnight only closed loop control (5 consecutive overnights) includes Module 1 and 3 (n=5-7).

ELIGIBILITY:
Inclusion Criteria:

1. ≥21 and <65 years old.
2. Clinical diagnosis of type 1 diabetes mellitus. For an individual to be enrolled at least one criterion from each list must be met.

   o Criteria for documented hyperglycemia (at least 1 must be met): i. Fasting glucose ≥126 mg/dL - confirmed ii. Two-hour Oral Glucose Tolerance Test glucose ≥200 mg/dL - confirmed iii. Hemoglobin A1C (HbA1c) ≥6.5% documented - confirmed iv. Random glucose ≥200 mg/dL with symptoms v. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes

   o Criteria for requiring insulin at diagnosis (1 must be met): i. Participant required insulin at diagnosis and continually thereafter ii. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually iii. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 1 year.
4. Familiarity with a bolus calculator with the current insulin pump with pre-defined parameters for carbohydrate ratio, insulin sensitivity factor (ISF), target glucose and active insulin.
5. HbA1c <9% as measured with DCA2000 or equivalent device.
6. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females).
7. Demonstration of proper mental status and cognition for the study.
8. Willingness to avoid consumption of acetaminophen-containing products 24 hours prior to and during CGM use.
9. Ability to access the Internet and upload CGM data via the company software during the data collection period.
10. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study.

Exclusion Criteria

1. Severe hypoglycemia resulting in seizure, loss of consciousness, or diabetic ketoacidosis within the 12 months prior to enrollment.
2. Pregnancy; breast feeding, or intention of becoming pregnant.
3. Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg).
4. Conditions which may increase the risks associated with possible hypoglycemia, such as any active cardiac disorder/arrhythmia, uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, uncontrolled adrenal insufficiency, neurologic disease or atrial fibrillation.
5. Self-reported hypoglycemia unawareness.
6. History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans.
7. Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the Continuous Glucose Monitor (CGM) (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants).
8. Anticoagulant therapy other than aspirin.
9. Oral steroids.
10. Subjects currently taking Amylin.
11. Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study sessions.
12. Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment).
13. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
14. Known current or recent alcohol or drug abuse.
15. Medical conditions that would make operating a CGM, the Diabetes Assistant (DiAs) cell phone or insulin pump difficult (e.g. blindness, severe arthritis, immobility).
16. Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, and cellulitis).
17. In adherence with the One Touch Ultra 2 User Guide that may be used in the experimental session and overnight during substudy, subjects with hematocrit levels less than 30% and above 55% will be excluded.
18. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase

    ≥three times the upper reference limit.
19. Impaired renal function measured as creatinine >1.2 times above the upper limit of normal.
20. Uncontrolled microvascular (diabetic) complications, such as current proliferative diabetic retinopathy or macular edema, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment.
21. Active gastroparesis requiring current medical therapy.
22. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study.
23. Uncontrolled thyroid disease.
24. Known bleeding diathesis or dyscrasia.
25. Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor.
26. Active enrollment in another treatment clinical trial. Observational trials may be permitted at the discretion of the study physician.
27. Use of anti-diabetic agents other than continuous subcutaneous insulin infusion (CSII) including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, Dipeptidyl peptidase-4 inhibitors, glucagon- like peptide 1 agonists, and alpha-glucosidase inhibitors
28. Unwillingness to use an approved form of birth control during this study by a sexually active female participant.
29. Subjects with basal rates less than 0.01U/hr.

RESTRICTIONS ON USE OF OTHER DRUGS OR TREATMENTS

1. Use of anti-diabetic agents other than CSII including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, Dipeptidyl peptidase-4 inhibitors, glucagon- like peptide 1 agonists, and alpha-glucosidase inhibitors.
2. Acetaminophen will be restricted starting 24 hours prior to CGM use.
3. Medications that block symptoms of hypoglycemia, including but not limited to beta blockers.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Brown SA, Kovatchev BP, Breton MD, Anderson SM, Keith-Hynes P, Patek SD, Jiang B, Ben Brahim N, Vereshchetin P, Bruttomesso D, Avogaro A, Del Favero S, Boscari F, Galasso S, Visentin R, Monaro M, Cobelli C. Multinight "bedside" closed-loop control for patients with type 1 diabetes. Diabetes Technol Ther. 2015 Mar;17(3):203-9. doi: 10.1089/dia.2014.0259. Epub 2015 Jan 16. PMID 25594434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Type 1 Diabetes recruited from medical clinics or local community.
Pre-assignment Details: This was a cross-over study in which subjects were assigned to either Overnight Closed-Loop Control (CLC) or Sensor-Augmented Pump Therapy (SAP) sessions first following training sessions.
  The additional AAA Control portion of the trial was not completed following pilot studies that indicated overnight closed-loop control to be preferable. Therefore the planned N=36 participants were not enrolled and no data was collected in the AAA Control 40hr portion of the trial.
Groups:
- Overnight CLC Control Followed by SAP: Participants had an CLC experimental session of 5 consecutive nights of closed loop control which was supervised in an outpatient setting. During the SAP control session, subjects were at home for a week using their home or study insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.
- SAP Followed by Overnight CLC: During the SAP control session, subjects were at home for a week using their home or study insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.Participants had an CLC experimental session of 5 consecutive nights of closed loop control which was supervised in an outpatient setting.
Period: First Phase (Overnight CLC or SAP)
Arm/Group | Overnight CLC Control Followed by SAP | SAP Followed by Overnight CLC
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Phase (SAP or Overnight CLC)
Arm/Group | Overnight CLC Control Followed by SAP | SAP Followed by Overnight CLC
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross-over trial with 10 participants total.
Groups:
- All Participants: Overnight CLC Control vs CGM + Insulin Pump at Home: Subjects had an Experimental session of 5 consecutive nights of closed loop control which was supervised. During the Control session, subjects will be at home using their home insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.
  The active comparator for subjects participating in 5 consecutive nights of closed loop control will be the sensor-augmented pump therapy at home in which the subject will be on their home insulin pump and using a CGM per their usual care.
Arm/Group | All Participants: Overnight CLC Control vs CGM + Insulin Pump at Home
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Cross-over trial with 10 participants total.
  years | 46.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5
  Italy | 5

OUTCOME MEASURES:

1. Primary Outcome: Time in Range Overnight
Description: For subjects participating in consecutive overnight control, will assess time in range (80-140mg/dL) overnight in closed loop control compared to sensor-augmented pump therapy.
Time Frame: 5 consecutive nights
Population: Cross-over trial with 10 participants total.
Measure: Mean (Inter-Quartile Range); unit: % time in range
Groups:
- Overnight Closed-Loop Control (CLC): Participants had an CLC experimental session of 5 consecutive nights of closed loop control (23:00 to 07:00) which was supervised in an outpatient setting.
- Sensor Augmented Pump Therapy (SAP): During the SAP control session, subjects were at home for a week using their home or study insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.
Arm/Group | Overnight Closed-Loop Control (CLC) | Sensor Augmented Pump Therapy (SAP)
Number analyzed (Participants) | 10 | 10
% time in range | 54.5 [36.5 to 74.7] | 32.2 [7.8 to 54.7]
Statistical Analysis 1: Comparison: Overnight Closed-Loop Control (CLC) vs Sensor Augmented Pump Therapy (SAP); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Evaluating the Risk for Hypoglycemia as Measured by the Low Blood Glucose Index
Description: A secondary goal of the cross-over trial is to evaluate the ability of the CLC to prevent hypoglycemia with the outcome measure of Low Blood Glucose Index. Low blood glucose index by CGM with higher index indicating higher risk of hypoglycemia. Values <1 suggest minimal risk (there is no maximum score). Index of risk of low blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale. The calculation of LBGI uses all available CGM values during the 5 consecutive nights of study to create one index. For the SAP group, the mean value lies outside the interquartile range due to outlying values that contribute to increasing the mean.
Time Frame: 5 consecutive nights
Measure: Mean (Inter-Quartile Range); unit: index score
Groups:
- Overnight CLC: Participants had an CLC experimental session of 5 consecutive nights of closed loop control (23:00 to 07:00) which was supervised in an outpatient setting.
- Sensor-Augmented Pump Therapy (SAP): During the Control Admission, subjects will use their home or study insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.
Arm/Group | Overnight CLC | Sensor-Augmented Pump Therapy (SAP)
Number analyzed (Participants) | 10 | 10
index score | 0.65 [0.02 to 0.84] | 1.05 [0 to 0.96]

3. Secondary Outcome: Time Within Target Range
Description: Closed loop control will improve the time spent within the target range of 70-180 mg/dl (computed from retrofitted CGM data).
Time Frame: 5 consecutive nights
Measure: Mean (Inter-Quartile Range); unit: % time in range
Groups:
- Overnight CLC: During the experimental CLC control sessions, participants stayed overnight at a supervised settling wearing the study insulin pump and two CGMs. Participants started the experimental system in pump only mode at 20:00 and at 23:00 switched to CLC mode overnight until 07:00. This session duration was 5 consecutive nights.
- Sensor-Augmented Pump Therapy (SAP): During the Control session, subjects will be at home and use their home or study insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.
Arm/Group | Overnight CLC | Sensor-Augmented Pump Therapy (SAP)
Number analyzed (Participants) | 10 | 10
% time in range | 85.4 [71.6 to 100] | 59.1 [30.2 to 100]

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected during the duration of the trial (consent through final study visit)
Groups:
- Overnight CLC: Participants had an Experimental session of 5 consecutive nights of closed loop control which was supervised.
- Sensor-Augmented Pump Therapy (SAP): During the Control session, subjects will be at home using their home or study insulin pump along with a continuous glucose monitor receiver without running any specialized mathematical equations.
Arm/Group | Overnight CLC | Sensor-Augmented Pump Therapy (SAP)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes